CLINICAL TRIAL: NCT05225168
Title: Comparison of Minisling Suburethral Sling Use and Laparoscopic Buch Colposuspension Application in Terms of Surgical Efficacy and Side Effects in True Stress Urinary Incontinence Surgery
Brief Title: Comparison of Minisling Suburethral Sling and Laparoscopic Buch Colposuspension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gamze Nur Cimilli Şenocak, assistant professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/284
Record Dates: First submitted 2022-01-26; First posted 2022-02-04 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Genuine Stress Incontinence
Keywords: Genuine Stress Incontinence; minisling; laparoscopic burch
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic burch colposuspension group (Active Comparator): this group will only have laparoscopic burch colposuspension
  Interventions: Procedure: laparoscopic burch colposuspension operation
- Minisling Suburethral Sling group (Active Comparator): this group will only have Minisling Suburethral Sling
  Interventions: Procedure: minisling suburethral sling

INTERVENTIONS:
Procedure: laparoscopic burch colposuspension operation — By pushing the urethra medially, two sutures are placed on the bladder at trigon level and midurethral and suspended on the bilateral iliopectineal ligament and colposuspension is supplied.
  Other Names: minisling suburethral sling
  Arms: laparoscopic burch colposuspension group
Procedure: minisling suburethral sling — A vertical vaginal incision is made 1 cm below the external urethral meatus. It is followed by minimal vaginal dissection from the inferior portion of the ascending ramus of the ischiopubic bone to the obturator muscle. The arms of the mesh are fixed on both sides of the obturator internus muscle with the help of a trocar. After leaving a 1-2 mm gap between the mesh and the urethra, the vaginal wall is closed by suturing.
  Arms: Minisling Suburethral Sling group

SUMMARY:
When the studies in the literature including the mini-sling procedure and the laparoscopic buch colposuspension procedure are examined, it is seen that both methods are successful in the surgical treatment of stress urinary incontinence (SUI), but there is no study in which both procedures have been found to be superior to each other in terms of efficacy and safety. The aim of this study is to compare the minisling suburethral sling and laparoscopic buch colposuspension application in terms of efficacy and side effects in patients who will undergo surgical treatment due to genuine SUI.

DETAILED DESCRIPTION:
When the studies in the literature including the mini-sling procedure and the laparoscopic buch colposuspension procedure are examined, it is seen that both methods are successful in the surgical treatment of stress urinery incontinence (SUI), but there is no study in which both procedures have been found to be superior to each other in terms of efficacy and safety. The aim of this study is to compare the minisling suburethral sling and laparoscopic buch colposuspension application in terms of efficacy and side effects in patients who will undergo surgical treatment due to genuine SUI. Investigators planned to measure patients' Kings Health Questionary and Prolapse Quality of Life test at first and 6 months after the surgery and to determine how the operation affects the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. To be between the ages of 18-80
2. Isolated genuine stress incontinence or accompanying pelvic organ prolapse
3. Having accepted surgery for stress urinary incontinence -

Exclusion Criteria:

* 1. Previously undergo pelvic organ prolapse surgery 2. Having a chronic lung disease such as asthma or Chronic obstructive pulmonary disease (COPD) 3. Having juvenile diabetes mellitus 4. History of gynecological cancer 5. Mesh allergy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-08-06 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
urinary stress test for evaluating objective cure | changes in urodynamics test at postoperative first and the 6th month
  In the postoperative period, urodynamics test will be determined at the 6th month and the absence of incontinence will be considered a cure.

SECONDARY OUTCOMES:
subjective continence | changes at postoperative first and the 6th month
  Patient satisfaction will be investigated by keeping a urinary diary and questioning the quality of life.
Prolapse quality of life (P-QoL) scale | changes at postoperative first and the 6th month
  Patients will be evaluated with the prolapse quality of life (P-QoL) scale. In this scale, the questions are rated 1 to 4, and as the total score increases, the quality of life decreases.
King's Health Questionnaire | changes at postoperative first and the 6th month
  Patients will be evaluated with the King's Health Questionnaire
Female sexual function scale (FSFI) | changes at postoperative first and the 6th month
  Patients will be evaluated with the Female sexual function scale (FSFI). In this scale, the questions are rated 0 to 5, and if the total score increases, it means the sexual life is better. A minimum of 2 and a maximum of 36 points can be obtained from this test.

CONTACTS AND LOCATIONS:
Overall Officials: Yakup Kumtepe, Study Director — Ataturk University; Yakup Kumtepe, Principal Investigator — Ataturk University
Locations (1):
- Gamze Nur Cimilli Senocak, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839